CLINICAL TRIAL: NCT01177007
Title: Intra-arterial Y-90 TheraSpheres for Hepatic Metastases From Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Jeff Geschwind, Professor of Radiology and Oncology, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J09150, NA_00035790; J09150 (Other: SKCCC Number)
Record Dates: First submitted 2010-08-02; First posted 2010-08-06 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Liver Neoplasms
Keywords: Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Neoplastic Processes; Pathologic Processes; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Adenocarcinoma; Neoplasms, Nerve Tissue; Liver Diseases; Neoplasms; Carcinoma; Colorectal Neoplasms; Neoplasm Metastasis; Carcinoma, Neuroendocrine; Liver Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases
MeSH Terms: conditions — Liver Neoplasms; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Neoplastic Processes; Pathologic Processes; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Adenocarcinoma; Neoplasms, Nerve Tissue; Liver Diseases; Neoplasms; Carcinoma; Colorectal Neoplasms; Neoplasm Metastasis; Carcinoma, Neuroendocrine; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TheraSphere (Experimental)
  Interventions: Device: TheraSphere, Yttrium-90 glass Microspheres

INTERVENTIONS:
Device: TheraSphere, Yttrium-90 glass Microspheres — Patients with unilobar disease will receive 120 ± 10% Gy (dose may be lower if clinically indicated) of TheraSphere to the affected lobe. Patients presenting with bilobar disease will have their liver assessed and the lobe presenting the highest treatment priority will receive the first treatment of TheraSphere. Assigning priority of lobes to receive treatment is based on tumor bulk, associated clinical symptoms attributed to the tumor and technical/angiographic considerations. In patients with bilobar disease where the second lobe does not require immediate treatment, or in unilobar disease where tumors develop in the untreated lobe, additional TheraSphere treatment may be administered at any subsequent time. A treatment may consist of a single 120 ± 10% Gy infusion to a lobe, or, if angiography indicates the need, the 120 ± 10% Gy dose may be split into multiple infusions per lobe to ensure delivery of a total of 120 ± 10% Gy to each treated lobe.

SUMMARY:
This study is an open label prospective trial of TheraSphere treatment for patients who have liver metastases who have failed or are intolerant to other systemic or liver directed therapies. Patients will be treated with TheraSphere at doses of 120 ± 10% Gy, and then followed for time to progression (TTP), safety, and overall survival.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older,
* Patients with a diagnosis of metastatic disease to the liver who have failed or are intolerant to other systemic or liver directed therapies.

A patient is considered to have failed to other systemic or liver-directed therapies when, in the opinion of the referring physician, the patient has progression of disease after receiving standard approved therapies. Specifically, if a patient has failed first line chemotherapy (or the standard approved therapies for that particular solid tumor), in the time period designed to assess that particular regimen (at least 30 days), then they may be enrolled into this protocol.

A patient is intolerant to other systemic or liver-directed therapies when, in the opinion of the referring physician, for example, the patient is unable to tolerate appropriate chemotherapy, when the patient had residual toxicity from previous therapies (e.g. neuropathy from oxaliplatin), or when the patient's performance status is such that treatment with systemic therapies would result in excessive toxicity.

* Liver metastases are unresectable
* Target tumors should be measurable using standard imaging techniques
* Tumor replacement ≤ 70% of total liver volume based on visual estimation by the Investigator
* Tumors are hypervascular based on visual estimation by the Investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2
* At least one month has elapsed since most recent prior cancer therapy with the following exceptions

  * Patients who are receiving Sandostatin for treatment of Neuroendocrine cancer may be enrolled and continue their Sandostatin treatment.
  * Patients receiving anti-oestrogen therapy for breast cancer may continue their treatment if therapy was initiated greater than 30 days prior to TheraSphere treatment.
  * Chemotherapy may continue if there is evidence of progression, in the liver, on treatment providing there is no change in the therapy in the 1 month prior to TheraSphere treatment and any immediate chemotherapeutic toxicity that will complicate TheraSphere treatment is resolved. In this case, the chemotherapy may continue because it is continuing to control the extrahepatic disease.
* Patient is willing to participate in the study and has signed the study informed consent

Exclusion Criteria

* At risk of hepatic or renal failure, as indicated by any of the following pre-treatment laboratory and clinical findings within 28 days of treatment:

  * Serum creatinine > 2.0 mg/dL, unless on dialysis
  * Serum total bilirubin ≥ 2.0 mg/dL
  * Albumin < 2.0 g/dL
  * Any history of hepatic encephalopathy
* Contraindications to angiography and selective visceral catheterization that may include, but are not limited to, the following:

  * Any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agents (e.g., closure device)
  * Severe peripheral vascular disease precluding catheterization
  * History of severe allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically.
* Severe liver dysfunction or presentation of pulmonary insufficiency or a clinically evident history of chronic obstructive pulmonary disease
* Cirrhosis or portal hypertension
* Previous external beam radiation treatment to the liver
* Any intervention for, or compromise of the Ampulla of Vater
* Clinically evident ascites. (Note: A radiographic finding of trace ascites on imaging is acceptable).
* Any continuing complications of prior cancer therapy that have not improved or resolved prior to 21 days before the first treatment with TheraSphere (if the investigator determines that the continuing complication will compromise the safety of the patient following treatment with TheraSphere).
* In the judgment of the physician, significant life-threatening extrahepatic disease
* Concurrent enrollment in another clinical study
* Evidence on technetium-99m macroaggregated albumin (99mTc-MAA) scan that demonstrates lung shunting with a potential absorbed dose of radiation to the lungs >30 Gy. The 30 Gy limit is a cumulative limit over all infusions of TheraSphere.
* Evidence on technetium-99m macroaggregated albumin (99mTc-MAA) scan that demonstrates a potential for the deposition of microspheres to the gastrointestinal tract that cannot be corrected by placement of the catheter distal to collateral vessels or using standard angiographic techniques, such as coil embolization.
* A positive serum pregnancy test in women of childbearing potential
* In the Investigator's judgment, any co-morbid disease or condition or event (e.g., recent myocardial infarction) that would place the patient at undue risk, and that would preclude safe use of TheraSphere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Geschwind, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients diagnosed with unresectable hepatic metastases who have failed or were intolerant to at least one line of systemic chemotherapy or liver-directed therapy. Participants were enrolled at Johns Hopkins Hospital with the last patient completed in April 2015.
Groups:
- TheraSphere: TheraSphere, Yttrium-90 glass Microspheres: Patients with unilobar disease will receive 120 ± 10% Gy (dose may be lower if clinically indicated) of TheraSphere to the affected lobe. Patients presenting with bilobar disease will have their liver assessed and the lobe presenting the highest treatment priority will receive the first treatment of TheraSphere. Assigning priority of lobes to receive treatment is based on tumor bulk, associated clinical symptoms attributed to the tumor and technical/angiographic considerations. In patients with bilobar disease where the second lobe does not require immediate treatment, or in unilobar disease where tumors develop in the untreated lobe, additional TheraSphere treatment may be administered at any subsequent time
Period: Overall Study
Arm/Group | TheraSphere
Started | 50
Completed First Y90 Treatment (Patients completing this milestone were analyzed for survival, safety, and dose outcomes) | 50
Completed First Clinical and Imaging (Patients completing this milestones were assessed for image response outcomes) | 43
Completed (Patients who completed all 12 months on protocol.) | 12
Not Completed | 38
Not completed — Lost to Follow-up | 2
Not completed — Death | 4
Not completed — Entered hospice care | 5
Not completed — Required additional Y90 treatment | 6
Not completed — Change in treatment modality | 21

BASELINE CHARACTERISTICS:
Arm/Group | TheraSphere
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [25 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) of the Treated Lesion(s) According to RECIST Criteria
Description: This outcome was not assessed. Instead, the primary outcome of progression-free survival based on RECIST and EASL criteria was assessed and reported.
Time Frame: Evaluated 4 weeks following each TheraSpheres procedure, and at 2-3 month intervals thereafter.
Population: These data were not collected. See outcome measure #2.
Groups:
- TheraSphere: TheraSphere, Yttrium-90 glass Microspheres: Patients with unilobar disease will receive 120 ± 10% Gy (dose may be lower if clinically indicated) of TheraSphere to the affected lobe. Patients with bilobar disease will have their liver assessed and the lobe presenting the highest treatment priority will receive the first treatment of TheraSphere. Assigning priority of lobes to receive treatment is based on tumor bulk, associated clinical symptoms attributed to the tumor and technical/angiographic considerations. In patients with bilobar disease where the second lobe does not require immediate treatment, or in unilobar disease where tumors develop in the untreated lobe, additional TheraSphere treatment may be administered at any subsequent time. A treatment may consist of a single 120 ± 10% Gy infusion to a lobe, or, if angiography indicates the need, the 120 ± 10% Gy dose may be split into multiple infusions per lobe to ensure delivery of a total of 120 ± 10% Gy to each tre
Arm/Group | TheraSphere
Number analyzed (Participants) | 0

2. Primary Outcome: Progression-free Survival (PFS) of the Treated Lesion(s) According to RECIST and EASL Criteria
Description: Progression-free survival was defined as the time from the date of Y-90 radioembolization to date of disease progression or latest follow-up. PFS was analyzed via Kaplan-Meier methodology with log-rank test using all 50 patients on study and stratified based on disease type. RECIST and EASL criteria were used to assess progression with kappa value for intermethod agreement of treatment responses of 0.9.
Time Frame: 2 years
Population: Median PFS for all subjects and stratified based on disease type.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TheraSphere
Number analyzed (Participants) | 50
months
  Median PFS for all disease types | 10.3 [7.6 to 13]
  Median PFS for CRC: number analyzed (Participants) | 12
  Median PFS for CRC | 22.0 [0 to 45.6]
  Median PFS for NE: number analyzed (Participants) | 26
  Median PFS for NE | 9.5 [2.4 to 16.6]
  Median PFS for non-CRC/non-NE: number analyzed (Participants) | 12
  Median PFS for non-CRC/non-NE | 15.8 [2.8 to 28.7]

3. Secondary Outcome: Time to Progression (TTP) of the Treated Lesion(s) According to EASL Criteria
Description: as for outcome 1
Time Frame: Evaluated 4 weeks following each TheraSpheres procedure, and at 2-3 month intervals thereafter.
Population: Analysis for TTP was not performed. In lieu of TTP, the PFS based on RECIST and EASL criteria was analyzed.
Groups:
- TheraSphere: TheraSphere, Yttrium-90 glass Microspheres: Patients with unilobar disease will receive 120 ± 10% Gy (dose may be lower if clinically indicated) of TheraSphere to the affected lobe. Patients presenting with bilobar disease will have their liver assessed and the lobe presenting the highest treatment priority will receive the first treatment of TheraSphere. Assigning priority of lobes to receive treatment is based on tumor bulk, associated clinical symptoms attributed to the tumor and technical/angiographic considerations. In patients with bilobar disease where the second lobe does not require immediate treatment, or in unilobar disease where tumors develop in the untreated lobe, additional TheraSphere treatment may be administered at any subsequent time. A treatment may consist of a single 120 ± 10% Gy infusion to a lobe, or, if angiography indicates, the 120 ± 10% Gy dose may be split into multiple infusions per lobe to ensure delivery of a total of 120 ± 10% Gy to each treated lob
Arm/Group | TheraSphere
Number analyzed (Participants) | 0

4. Secondary Outcome: Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST) v1.0
Description: Efficacy as assessed by radiographic tumor response using RECIST criteria at baseline, at 4 weeks post treatment, and subsequent 3 month intervals.
  Complete Response (CR): Disappearance of all lesions targeted by Y90 Partial Response (PR): At least 30% decrease in the sum of longest diameter (LD) of lesions targeted by Y90 Progressive Disease (PD): At least 20% increase in sum of LD of lesions targeted by Y90 Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD.
Time Frame: 12 months
Population: RECIST for all applicable patients (n=43) were analyzed and also stratified based on disease type: CRC (n=9); NE (n=22); and non-CRC/non-NE (n=12).
Measure: Count of Participants; unit: Participants
Arm/Group | TheraSphere
Number analyzed (Participants) | 43
Participants
  All disease types: Complete Response (CR) | 11
  All disease types: Partial Response (PR) | 9
  All disease types: Stable Disease (SD) | 11
  All disease types: Progressive Disease (PD) | 12
  Colorectal cancer only: number analyzed (Participants) | 9
  Colorectal cancer only: Complete Response (CR) | 1
  Colorectal cancer only: Partial Response (PR) | 3
  Colorectal cancer only: Stable Disease (SD) | 2
  Colorectal cancer only: Progressive Disease (PD) | 3
  Neuroendocrine only: number analyzed (Participants) | 22
  Neuroendocrine only: Complete Response (CR) | 7
  Neuroendocrine only: Partial Response (PR) | 4
  Neuroendocrine only: Stable Disease (SD) | 6
  Neuroendocrine only: Progressive Disease (PD) | 5
  Non-CRC/Non-NE: number analyzed (Participants) | 12
  Non-CRC/Non-NE: Complete Response (CR) | 3
  Non-CRC/Non-NE: Partial Response (PR) | 2
  Non-CRC/Non-NE: Stable Disease (SD) | 3
  Non-CRC/Non-NE: Progressive Disease (PD) | 4

5. Secondary Outcome: Tumor Response by the European Association for the Study of the Liver (EASL) Criteria
Description: Efficacy as assessed by radiographic tumor response using EASL criteria at baseline up to 12 months post treatment.
  Complete Response (CR): Achieving 100% tumor necrosis of targeted lesions Partial Response (PR): Demonstrating greater than 50% tumor necrosis in targeted lesions Progressive Disease (PD): Reappearance of or increased tumor enhancement greater than 25% in targeted lesions Stable Disease (SD): Not meeting requirements for CR or PR and not demonstrating evidence of progression in targeted lesions.
Time Frame: 12 months
Population: RECIST for all applicable patients (n=43) were analyzed and also stratified based on disease type: CRC (n=9); NE (n=22); and non-CRC/non-NE (n=12). 7 out of the 50 patients were not analyzed due to lack of follow-up imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | TheraSphere
Number analyzed (Participants) | 43
Participants
  All disease types: Complete Response (CR) | 11
  All disease types: Partial Response (PR) | 9
  All disease types: Stable Disease (SD) | 10
  All disease types: Progressive Disease (PD) | 13
  Colorectal cancer only: number analyzed (Participants) | 9
  Colorectal cancer only: Complete Response (CR) | 1
  Colorectal cancer only: Partial Response (PR) | 2
  Colorectal cancer only: Stable Disease (SD) | 3
  Colorectal cancer only: Progressive Disease (PD) | 3
  Neuroendocrine only: number analyzed (Participants) | 22
  Neuroendocrine only: Complete Response (CR) | 7
  Neuroendocrine only: Partial Response (PR) | 5
  Neuroendocrine only: Stable Disease (SD) | 4
  Neuroendocrine only: Progressive Disease (PD) | 6
  Non-CRC/Non-NE: number analyzed (Participants) | 12
  Non-CRC/Non-NE: Complete Response (CR) | 3
  Non-CRC/Non-NE: Partial Response (PR) | 2
  Non-CRC/Non-NE: Stable Disease (SD) | 3
  Non-CRC/Non-NE: Progressive Disease (PD) | 4

6. Secondary Outcome: Overall Survival (OS)
Description: Measured from the date corresponding to initiation of therapy until the date of death due to any cause. At the time of registration, the outcome measure was entered in clinicaltrials.gov as "open-ended". Overall survival was analyzed via Kaplan-Meier methodology with log-rank test using all 50 patients on study and stratified based on disease type.
Time Frame: Median follow-up time was 11.41 months (CI: 1.5-33.7)
Population: Median OS for all patients (n=50) were analyzed and also stratified based on disease type: CRC (n=12); NE (n=26); and non-CRC/non-NE (n=12).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TheraSphere
Number analyzed (Participants) | 50
months
  Median OS for all disease types | 11.7 [10.6 to 12.8]
  Median OS for CRC: number analyzed (Participants) | 12
  Median OS for CRC | 11.9 [10.9 to 12.8]
  Median OS for NE: number analyzed (Participants) | 26
  Median OS for NE | 7.6 [0 to 15.9]
  Median OS for non-CRC/non-NE: number analyzed (Participants) | 12
  Median OS for non-CRC/non-NE | 15.8 [10.9 to 20.9]

7. Secondary Outcome: Overall Survival (OS) Rate at 2 Years
Description: Measured from the date corresponding to initiation of therapy until the date of death due to any cause. At the time of registration, the outcome measure was entered in clinicaltrials.gov as "open-ended". At the time of results reporting, this outcome was presented as "Up to 2 years". Overall survival was analyzed via Kaplan-Meier methodology with log-rank test using all 50 patients on study and stratified based on disease type. 2-year OS rates were also stratified based on tumor burden.
Time Frame: Up to 2 years
Population: 2-year OS rate for all patients (n=50) were analyzed and also stratified based on tumor burden: Patients with tumor burden of 25% or less (n=34) and patients with tumor burden greater than 25% (n=16).
Measure: Number; unit: percentage of participants
Arm/Group | TheraSphere
Number analyzed (Participants) | 50
percentage of participants
  OS rate for all patients | 22
  OS rate for tumor burden greater than 25%: number analyzed (Participants) | 16
  OS rate for tumor burden greater than 25% | 0
  OS rate for tumor burden 25% or less: number analyzed (Participants) | 34
  OS rate for tumor burden 25% or less | 36

8. Secondary Outcome: Safety as Graded by CTCAE Version 3.0
Description: Clinical and biochemical toxicity that were assessed as at least possibly related to treatment were recorded from the day of treatment until protocol exit or death. Toxicities were graded by the Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Time Frame: 12 months
Population: 50 participants were assessed for adverse events, with a total of 207 adverse events reported. Two patients had grade 5 toxicities (grade 5 cholecystitis and death), which were attributed to disease progression and were not device-related.
Measure: Number; unit: adverse events
Units Other Than Participants: Adverse Events
Arm/Group | TheraSphere
Number analyzed (Participants) | 50
Number analyzed (Adverse Events) | 207
adverse events
  Elevated alkaline phosphatase | 21
  Elevated ALT | 13
  Elevated AST | 11
  Lymphocyte depression (asymptomatic) | 23
  Fatigue | 33
  Fever | 8
  Nausea | 19
  Heartburn | 6
  Vomiting | 6
  Pain | 23
  Decreased albumin | 4
  Elevated bilirubin | 3
  Anorexia | 11
  Weight loss | 13
  Constipation | 7
  Muscle pain | 1
  Cholecystitis | 1
  Death (disease progression) | 1
  Allergic reaction (contrast media) | 1
  Thrombosis/embolism (vascular access) | 1
  Liver failure | 1

9. Secondary Outcome: Mean Radiation Dose Delivered to Total Liver
Description: Therasphere dose calculation was performed using positron emission tomography-computed tomography (PET/CT) and single-photon emission computed tomography (SPECT) imaging post-procedure to estimate the actual delivered dose of Theraspheres to the liver.
Time Frame: 24 hours
Population: Mean radiation doses were calculated for the total cohort of participants and also stratified according to disease type - colorectal cancer, neuroendocrine, and non-CRC/non-NE.
Measure: Mean (Standard Deviation); unit: Gray
Arm/Group | TheraSphere
Number analyzed (Participants) | 50
Gray
  Mean radiation dose for all patients | 112.13 (13.56)
  Mean dosing for CRC: number analyzed (Participants) | 12
  Mean dosing for CRC | 115.57 (10.97)
  Mean dosing for NE: number analyzed (Participants) | 26
  Mean dosing for NE | 109.41 (13.08)
  Mean dosing for non-CRC/non-NE: number analyzed (Participants) | 12
  Mean dosing for non-CRC/non-NE | 115.18 (16.37)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | TheraSphere
All-Cause Mortality (participants affected / at risk) | 4/50
Serious Adverse Events (participants affected / at risk) | 14/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TheraSphere (N=50)
Death (disease progression) (General disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Brain surgery for metastatic disease (Surgical and medical procedures) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Failure to thrive (Investigations) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Cardiac infarction (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Acetaminophen overdose (Investigations) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TheraSphere (N=50)
Distension/bloating, abdominal (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 19 (21)
Edema: trunk (General disorders) | 1 (1)
Lymphopenia (Investigations) | 35 (54)
Diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2)
Neutropenia (Investigations) | 2 (2)
Elevated AST (Investigations) | 25 (31)
Elevated ALT (Investigations) | 15 (16)
Anemia (Blood and lymphatic system disorders) | 11 (12)
Acid reflux (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 21 (23)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (13)
Elevated alkaline phosphatase (Investigations) | 29 (32)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (17)
Confusion (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 12 (15)
Depression (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Fatigue (General disorders) | 35 (49)
Fever (General disorders) | 12 (14)
Hyperbilirubinemia (Investigations) | 10 (11)
Elevated INR (Investigations) | 5 (5)
Concentration impairment (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 26 (37)
Neuropathy (Nervous system disorders) | 6 (7)
Headache (Nervous system disorders) | 8 (11)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Leukopenia (Investigations) | 14 (17)
Night sweat (Vascular disorders) | 8 (12)
Thrombocytopenia (Investigations) | 9 (10)
Vomiting (Gastrointestinal disorders) | 11 (11)
Elevated creatinine (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Weight gain (Investigations) | 7 (9)
Weight loss (Investigations) | 14 (18)
Chills (General disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Hypercalcemia (Investigations) | 1 (1)
Hyperglycemia (Investigations) | 17 (23)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 11 (11)
Pain - general (General disorders) | 4 (4)
Pain - site of incision (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Chest pain - non-cardiac (General disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain - stomach (Gastrointestinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Lower extremity edema (General disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Visual changes (Eye disorders) | 2 (2)
Hot flash (Vascular disorders) | 3 (3)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes